CLINICAL TRIAL: NCT06585878
Title: Study on the Efficacy and Safety of Vorolanib Combined With Cadonilimab in the Treatment of Untreated Advanced RCC Patients
Brief Title: A Prospective Registry Study of Stereotactic Ablative Radiotherapy (SABR) for Oligometastatic/Oligometastatic Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiongjun Ye, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4712
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Renal Cell Carcinoma; RCC; Kidney Cancer
Keywords: Renal Cell Carcinoma; Stereotactic Ablative Radiotherapy (SABR); Systemic Treatment; Toxicity; Curative Effect
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): SBRT radiotherapy for all lesions/all metastatic lesions
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — Without altering the patients' systemic treatment plans, patients who meet the inclusion criteria after MDT discussion will receive SBRT radiotherapy for all lesions/all metastatic lesions based on the guideline-recommended medications. The radiotherapy plan is based on the SABR-COMET protocol and Timmerman's constraints.

SUMMARY:
Study the efficacy and toxicity of SABR treatment for oligometastatic/oligoprogressive renal cell carcinoma; investigate the effectiveness and safety of SABR combined with targeted immunotherapy; conduct stratified analysis to identify the optimal beneficiary population; establish a biobank to screen for biomarkers; and use radiomics analysis to identify characteristics of sensitive populations.

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, registry-based trial that aims to enroll 60 patients with renal cancer who will be diagnosed and treated at our hospital between May 2024 and May 2026. Without altering the patients' systemic treatment plans, those who meet the inclusion criteria after MDT discussion will receive SBRT (Stereotactic Body Radiation Therapy) for all lesions/all metastatic lesions in addition to the guideline-recommended medications. The radiotherapy plan is based on the SABR-COMET protocol and Timmerman's constraints. Patient data will be collected, including general clinical information, toxicity assessments during treatment and in the acute phase, detailed imaging data, regular assessments of pain and quality of life, and evaluations of late radiation therapy responses.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients with newly diagnosed M1 renal cancer or those with oligoprogression during systemic therapy, with no restrictions on the location or number of metastatic sites, but all metastatic sites must be evaluated by the radiation oncology department as safely able to receive a radical radiation dose (α/β value of 3, EQD2 ≥ 70Gy).

  2: Age ≥ 18 years. 3: ECOG score of 0-3. 4: Confirmed renal malignancy by pathology or imaging examination, with no subtype restrictions.

  5: Presence of evaluable lesions. 6: Patients with spinal cord compression or significant brain metastasis edema requiring surgical decompression can be enrolled after evaluation by the radiation oncology department if the aforementioned dose can be safely administered post-decompression.

  7: Able to tolerate radiation therapy and standard systemic therapy (targeted therapy or targeted immunotherapy combination).

  8: Expected survival > 6 months. 9: Able to sign the informed consent form. 10: Has conditions for follow-up.

Exclusion Criteria:

* 1: Patients with other comorbidities that prevent the use or tolerance of targeted immunotherapy drugs, such as targeted immunotherapy drug allergies, active bleeding, ulcers, intestinal perforation, intestinal obstruction, uncontrolled hypertension, grade III-IV cardiac dysfunction (NYHA criteria), severe hepatic and renal insufficiency (grade IV), etc.

  2: Patients with other comorbidities that prevent tolerance of radiation therapy.

  3: Complete response to first-line drug therapy (i.e., no treatable targets for SABR).

  4: Previous history of radiation therapy to the same site. 5: Pregnant or lactating women. 6: Patients with other severe medical comorbidities that prevent participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Through study completion, an average of 2 year
  K-M survival curves

SECONDARY OUTCOMES:
2 Years Progression-Free Surial | For all the patients, the time from the index of treatment to 2 years
  K-M survival curves
2 Years Overall Survival | For all the patients, the time from the index of treatment to 2 years
  K-M survival curves
Life Quality Score | Through study completion, an average of 2 year，at each follow-up visit，once a month.
  TESS score, scores range from 0 to 60, with higher values indicating better quality of life.
Pain Score | Through study completion, an average of 2 year，at each follow-up visit，once a month.
  VRS grading system, a five-point scale is used, with higher scores indicating more severe perceived pain.
Acute Toxicity | Through study completion, an average of 2 year，at each follow-up visit，once a month.
  Adopt CTCAE5.0 standard, a six-point scale is used, 0 to 5 scale, with higher scores indicating more severe adverse reaction.

IPD SHARING:
Plan to Share IPD: No